CLINICAL TRIAL: NCT05505617
Title: Comparison Between Two Commercially Available Devices to Measure Nitric Oxide Lung Diffusing Capacity in Systemic Sclerosis: a Randomized Crossover Trial
Brief Title: Nitric Oxide Lung Diffusing Capacity in Systemic Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Holger Dressel (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Holger Dressel, Prof. Dr med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2022-00280
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Systemic Sclerosis
Keywords: nitric oxide; DLNO
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung diffusing capacity measurements: Participants will be randomly allocated to perform single-breath lung diffusing capacity measurements on both devises during a single study visit.
  Interventions: Other: Single-breath nitric oxide lung diffusing capacity measurements according to type of device in random order.

INTERVENTIONS:
Other: Single-breath nitric oxide lung diffusing capacity measurements according to type of device in random order. — Device: Jaeger Masterscreen TM (PFT Pro, Vyaire, Hoechberg, Germany)
  Device: HypAir Medisoft (Medisoft, Dinant, Belgium)

SUMMARY:
To date, two devices to measure nitric oxide lung diffusing capacity (DLNO) are commercially available in Europe. Previous research has shown systematic between-device differences in lung diffusing capacity outcomes in healthy people (Radtke et al. ERJ Open Res. 2021 Sep 13;7(3)). The extent and magnitude of between-device differences in people with lung function impairment and ventilation inhomogeneities is unknown.

DETAILED DESCRIPTION:
The aim of this project is to compare two commercially available devices that measure lung diffusing capacity for nitric oxide (DLNO) in people with systemic sclerosis and proven interstitial lung disease.

1. "MasterScreenTM" (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany
2. "HypAir" ("HA", Medisoft, Dinant, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of systemic sclerosis by American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR1) criteria (≥ 9 points)
* Interstitial lung disease proven with high-resolution computed tomography (HRCT)
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Unstable clinical condition affecting lung function testing (i.e., major hemoptoe/-tysis or pneumothorax within the last 3 months, acute respiratory tract infection in the past two weeks), others according to the assessment of the treating physician
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with systemic sclerosis and computed tomography proven interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in nitric oxide lung diffusing capacity (DLNO in mL.min-1.mmHg-1) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).

SECONDARY OUTCOMES:
Difference in carbon monoxide lung diffusing capacity (DLCO in mL.min-1.mmHg-1) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in Alveolar volume (VA in L) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in the physiological rate of NO uptake from alveolar gas (KNO in mL.min.-1mmHg-1.L-1) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in the physiological rate of CO uptake from alveolar gas (KCO in mL.min.-1mmHg-1.L-1) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in the rate constant for NO removal from alveolar gas (κNO in s-1) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in the rate constant for CO removal from alveolar gas (κCO in s-1) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in change in fractional alveolar NO concentration (ΔFA NO in ppm) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in change in fractional alveolar CO concentration (ΔFA CO in %) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in breath-hold time (BHT in s) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for nitric oxide (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for nitric oxide (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for carbon monoxide (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for carbon monoxide (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for oxygen (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for oxygen (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for helium (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for helium (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).

CONTACTS AND LOCATIONS:
Overall Officials: Holger Dressel, Prof, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be made available upon publication in an open-access journal.

REFERENCES:
- [Background] Erratum: "Lung diffusing capacity for nitric oxide measured by two commercial devices: a randomised crossover comparison in healthy adults". Thomas Radtke, Quintin de Groot, Sarah R. Haile, Marion Maggi, Connie C.W. Hsia and Holger Dressel. ERJ Open Res 2021; 7: 00193-2021. ERJ Open Res. 2021 Sep 13;7(3):50193-2021. doi: 10.1183/23120541.50193-2021. eCollection 2021 Jul. PMID 34527728